CLINICAL TRIAL: NCT05807659
Title: Fractionated Busulfan Combined With Chidamide/Fludarabine/Cytarabine (ChiFAB) With Allogeneic Hematopoietic Stem-Cell Transplantation in Non-remission Myeloid Malignancies: a Phase II Study
Brief Title: Fractionated Busulfan Conditioning Regimen for Allo-HSCT in Non-remission Myeloid Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fra-Bu 1.0
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Myeloid Malignancies
Keywords: myeloid malignancies; allo-HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fractionated busulfan (Experimental): fractionated busulfan-based ChiFAB conditioning regimen: busulfan 3.2mg/kg d-13, -12, 1.6mg/kg d-6~-3, fludarabine 35mg/m2 d-6~-2 cytarabine 1g/m2,d-6~-2 chidamide 30mg d-13,-10,-6,-3
  Interventions: Drug: fractionated busulfan-based conditioning regimen

INTERVENTIONS:
Drug: fractionated busulfan-based conditioning regimen — Drug: Chidamide 30 mg oral twice weekly for 2 weeks Drug: Fludarabine 35 mg/m2 intravenously daily for 5 days in the 2nd week Drug: Cytarabine
  1 g/m2 intravenously for 5 days in the 2nd week Drug: Busulfan 3.2 mg/kg intravenously daily for 2 days in the 1st week, 1.6 mg/kg intravenously daily for 4 days in the 2nd week Procedure/Surgery: allogeneic hematopoietic stem cell transplantation

SUMMARY:
The goal of this single-arm phase II study is to test in patients with non-remission myeloid malignancies undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT). The main question it aims to answer are:

* The safety and efficacy of fractionated busulfan Combined With Chidamide/Fludarabine/Cytarabine(ChiFAB) conditioning regimen in increasing the overall survival rate in patients with non-remission myeloid malignancies after allo-HSCT.
* The efficacy of fractionated busulfan conditioning regimen in reducing the recurrence rate in patients with non-remission myeloid malignancies after allo-HSCT.

Participants will receive fractionated busulfan-based ChiFAB conditioning regimen (busulfan 3.2mg/kg d-13, -12, 1.6mg/kg d-6~-3, fludarabine 35mg/m2 d-6~-2, cytarabine 1g/m2,d-6~-2, chidamide 30mg d-13,-10,-6,-3) before allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 65 years old when signing the Informed Consent Form (ICF);
2. KPS score > 60 or ECOG score 0-2;
3. The expected survival period > 3 months;
4. Those who did not achieve complete remission after 2 or more chemotherapy regimens. The proportion of blasts on bone marrow smears before transplantation was ≥5%.
5. Those who have no central nervous system involvement or serious functional damage to important organs of the body;
6. Fully understand and be informed of this study and sign the ICF; willing to follow and have the ability to complete all test procedures;

Exclusion Criteria:

1. Serious basic diseases of important organs: such as myocardial infarction, chronic cardiac insufficiency, decompensated hepatic insufficiency, renal function, gastrointestinal insufficiency, etc.;
2. Uncontrolled active infection (including bacterial, fungal, or viral infection), and drug treatment is ineffective;
3. Participating in other clinical studies, or planning to start treatment in this study and less than 4 weeks before the end of treatment in the previous clinical study;
4. Combined with other malignant tumors and require treatment;
5. Pregnant or lactating females;
6. Patients with known history of human immunodeficiency virus (HIV) virus infection and/or acquired immunodeficiency syndrome;
7. Patients with active chronic hepatitis B or active hepatitis C;
8. History of prolonged QT syndrome;
9. Patients considered by other researchers to be unsuitable for this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival of this group of patients at the end of 2 year

SECONDARY OUTCOMES:
Non-relapse mortality (NRM) | 6 months
  Non-relapse mortality of this group of patients at the end of 6 months
Relapse rate | 2 years
  Relapse rate of this group of patients at the end of 2 year
Cumulative incidence of acute graft versus host disease (aGVHD) | Day +100
  Cumulative incidence of acute graft versus host disease (aGVHD) of this group of patients at day+100
Cumulative incidence of chronic graft versus host disease (cGVHD) | 2 years
  Cumulative incidence of chronic graft versus host disease (cGVHD) of this group of patients at the end of 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Release after the publication of results of this trial
Supporting Information: Study Protocol
Time Frame: after the publication of results of this trial